CLINICAL TRIAL: NCT03749629
Title: Comparative Effectiveness of Pharmacogenomics for Treatment of Depression
Acronym: CEPIO-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genetic Alliance (Other); Patient-Centered Outcomes Research Institute (Other); Vanderbilt University (Other); Montefiore Medical Center (Other); Louisiana State University Health Sciences Center in New Orleans (Other); Duke University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P002499
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; Pharmacogenomic testing
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Intervention Model Description: Investigators will prospectively randomize 400 participants with DSM-V major depressive disorder to best practice guidelines plus PGx- guided psychiatric treatment (n=200) or best practice guidelines alone (n=200) and follow them for one year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CANMAT + GeneSight Psychotropic Test guided tx (Active Comparator): Participant treatment will be guided by the Canadian Network for Mood and Anxiety Treatments (CANMAT) and the pharmacogenomic test GeneSight®. GeneSight® is a neuropsychiatric, combinatorial, PGx test that provides recommendations for psychotropic medications (antidepressants, mood stabilizers, hypnotics for insomnia, and antipsychotics) based on a patient's individual genetic profile.
  Interventions: Other: GeneSight Psychotropic test; Other: Canadian Network for Mood and Anxiety Treatment (CANMAT) Best Practice Guidelines
- CANMAT alone (Placebo Comparator): Participant treatment will be guided by the Canadian Network for Mood and Anxiety Treatments (CANMAT) alone.
  Interventions: Other: Canadian Network for Mood and Anxiety Treatment (CANMAT) Best Practice Guidelines

INTERVENTIONS:
Other: GeneSight Psychotropic test — GeneSight® Psychotropic powered by CPGx® technology, the only test for depression reimbursable by Medicaid and Medicare. GeneSight® is a neuropsychiatric, combinatorial, PGx test that provides recommendations for psychotropic medications (antidepressants, mood stabilizers, hypnotics for insomnia, and antipsychotics) based on a patient's individual genetic profile.
  Arms: CANMAT + GeneSight Psychotropic Test guided tx
Other: Canadian Network for Mood and Anxiety Treatment (CANMAT) Best Practice Guidelines — Guidelines for treatment

SUMMARY:
The overall goal of this study is to assess the effectiveness of a widely available and widely used combinatorial pharmacogenomic (PGx) test for the treatment of major depressive disorder. Pharmacogenomic tests use genetic information to guide medication treatment decisions. The tests inform clinicians and patients of potential gene-drug interactions by analyzing pharmacokinetic (PK) genes (how drugs are metabolized) as well as pharmacodynamic (PD) genes (how drugs work). While combinatorial PGx testing is attractive to clinicians, patients, healthcare systems, and insurers, limited data demonstrate that PGx testing will result in better outcomes compared to evidence-based guideline treatment. Therefore, the investigators will conduct a prospective randomized comparative effectiveness study of best practice guidelines plus combinatorial PGx-guided treatment versus best-practice guideline concordant treatment alone.

DETAILED DESCRIPTION:
Depressive disorders are the fourth leading cause of the burden of disease worldwide and is projected to be the first cause by 2030 1. According to the World Health Organization depression carries the greatest burden of disability among all mental and behavioral disorders. Specifically, depression accounts for 3.7% of all U.S. disability-adjusted life years and 8.3% of all U.S. years lived with disability. In 2014, it was estimated that 15.7 million adults in the United States had at least one major depressive episode in the past year and 43% people with severe depressive symptoms reported serious difficulties in work, home, and social activities 2. The current standard of care is based on trial-and-error of a multitude of medications; this approach often leads to patient and clinician frustration after each treatment failure (side effects or non-response) and can decrease compliance and engagement in treatment. One way to reduce this trial-and-error process, is to use pharmacogenomic (PGx) testing to guide medication treatment and increase the likelihood of response by reducing the number of ineffective medication trials.

Pharmacogenomics, the use of genetic information by patients, clinicians, and healthcare systems to match patients with pharmacologic treatments, is an important step towards precision/personalized medicine. Pharmacogenomics can make the practice of medicine more efficient by giving the right medications specifically to those who are most likely to benefit from them and to avoid giving the wrong medications to those who are most likely not to benefit based on each patient's individual genetic makeup. The PGx test for the treatment of depression is now commercially available and is reimbursable by insurance, including Medicaid and Medicare. A recent comprehensive overview of the state of PGx testing for depression, its promise, and limitations concluded that more research is needed in this rapidly-developing field3. Specifically, the gap is that while PGx-guided antidepressant treatment results in better outcomes compared to treatment as usual in tightly controlled clinical trials, it has not yet been tested in real world settings, nor has it been compared to best practice guidelines. It is less clear how well PGx tests make a difference in short and long-term patient-centered outcomes compared to guideline-concordant care of depression.

For this study, the investigators are collaborating with Assurex Health and their product GeneSight® Psychotropic powered by CPGx® technology, the only test for depression reimbursable by Medicaid and Medicare. GeneSight® is a neuropsychiatric, combinatorial, PGx test that provides recommendations for psychotropic medications (antidepressants, mood stabilizers, hypnotics for insomnia, and antipsychotics) based on a patient's individual genetic profile. The test combines pharmacokinetic (PK) metabolism genes (how drugs are metabolized) as well as pharmacodynamic (PD) genes (how drugs work) to predict dosing adjustments and response.

GeneSight® classifies medications based on the severity of the gene-drug interactions in color-coded categories: green "use as directed," yellow "moderate gene-drug interaction," and red "significant gene-drug interaction." The results are presented in a report which is easily understandable by patients and clinicians. Furthermore, GeneSight® addresses concerns reported by individuals in MoodNetwork: alleviating symptoms, identifying effective alternative treatments, reducing barriers to care/treatment, and using genetic studies to identify responders to treatment. This study answers questions that patients and clinicians care about and has the potential to improve outcomes.

Cogito, Inc. is the industry leader in the mobile sensing technology of mood. Cogito has developed a mobile phone application that assesses depression by tracking everyday usage of mobile phones, without the need to actively input data (e.g., rating depression). The application uses indicators such as phone call/text frequency or voice parameters to deduce depression severity. To date, this application has been tested in two studies: Defense Advanced Research Projects Agency (DARPA) funded a study in 73 patients with major depression and PTSD3, and a more recent NIMH funded study with 200 patients with major depression and bipolar disorder in collaboration with the MoodNetwork PPRN. The application is highly sensitive and specific in detecting depression. However, given the preliminary nature of these findings, the study investigators will use the Cogito platform as a secondary (more exploratory) outcome measure and the use of this application will be optional. The use of passive sensing technology has the advantage that it does not rely on patients' self-report and can be used for low cost longitudinal monitoring of patients for the changes in depression symptoms.

If a study clinician meets with one of their patients and determines that they may be eligible for the study, a member of the study staff (i.e. site PI, treating clinician, or research assistant) will describe the study to the patient and answer any questions. If the participant is interested, they will complete the consent form accessed via MoodNetwork.org. Patients will be offered to take home the Consent Form and call back if they wish to participate. If they decide to participate, they will contact the member of the research team and will be given the study website link to sign consent. Following their consent, participants will be prompted to complete questionnaires to determine study eligibility on MoodNetwork.org. If the patient is eligible for the study, they will be informed of the option to use the Cogito Companion mobile app and if they want to use it, they will be asked to download the mobile app (so that the study team can passively monitor any potential depressive symptoms throughout the course of the study) and they will be randomized to either the PGx-guided psychiatric treatment arm or the best practice guidelines arm. A member of study staff will then administer the PGx test (i.e., a buccal swab). If the participant is in the PGx-guided psychiatric treatment arm, the treating clinician will receive their results within two business days and contact the participant to inform them of the results and discuss any medication changes. If the participant is in the best practice guidelines arm, the treating clinician will not receive the PGx test results until after the follow-up phase (one year). The clinician, however, will still contact the patient to discuss medication changes (in line with the Canadian Network for Mood and Anxiety Treatments (CANMAT) guidelines instead of the GeneSite test results).

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Between the ages of 18-65
* Diagnosed with Major Depressive Disorder (assessed by the Composite International
* Diagnostic Interview Screening Scales (CIDI-SC))
* Currently Depressed (PHQ 9 ≥10)

Exclusion Criteria:

* Diagnosis of bipolar disorder or schizophrenia
* Patients posing a serious suicidal risk and/or in need of immediate hospitalization as judged by the treating clinician
* Has a general medical condition that is responsible for depressive symptoms or uses a medication responsible for depressive symptoms
* Any medical contraindications for participants to take study medications
* Patients with a history of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic or euthyroid for 6 months
* Patients with significant unstable medical condition; life threatening disease; hepatic insufficiency (3X Upper Limit of Normal (ULN) for AST and/or ALT); liver transplant recipient; cirrhosis of the liver; need for therapies that may obscure the results of treatment and/or of the study; malignancy (except basal cell carcinoma) and/or chemotherapy within 1 year prior to screening
* Patients with a history of gastric bypass surgery. (This exclusion depends on the type of gastric bypass surgery. Those that simply restrict the size of the stomach are acceptable.
* Those that alter the ability of the stomach/digestive lining to absorb nutrients are not. GeneSight is unable to account for absorption issues due to this reason at this time.)
* Patients who self-report to be pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Well-being as assessed by the World Health Organization Well-Being Index (WHO-5) | 1 year
  Hypothesis: Combinatorial PGx-guided treatment will be superior to best-practice guideline treatment to increase well-being The World Health Organization-5 Well-Being Index (WHO-5, primary outcome measure) is a brief 5-item self-report questionnaire consisting of positively-worded statements related to positive mood, vitality, and general interests over the prior two weeks. Item scores range from 0 (none of the time) to 5 (all of the time), resulting in a range of summary scores from 0 (poor well-being) to 25 (optimal well-being).

SECONDARY OUTCOMES:
Depression severity | 1 year
  Patient Health Questionnaire (PHQ-9)- The Patient Health Questionnaire-9 (PHQ-9) is a brief self-report instrument used to screen, diagnose, monitor, and measure the severity of depression. The first 8 questions incorporate DSM-IV diagnostic criteria as well as other major depressive symptoms, and Question 9 assesses for the presence and duration of suicidal ideation.
Necessary medication adjustments | 1 year
  Medication Recommendation Tracking Form (MRTF) Study clinicians will use this online medication tracking form that we have used in our previous large-scale, clinical trials conducted on the Bipolar Trials Network to record the dates of starting and stopping psychotropic medications as well as the reasons for discontinuation.
Functioning | 1 year
  Patient-Reported Outcomes Measurement Information System (PROMIS) Functioning Functioning will be measured via the PROMIS 29Ability to Participate in Social Roles and Activities" Index. This scale consists of 4 items that inquire about a person's ability to do leisure or family activities, perform usual work activities (including work at home), or engage in desired activities with friends in the past 7 days. Items are rated on a 5-point rating scale ranging from "Never" to "Always", resulting in a range of scores from "0" to "20", with "0" indicating maximum impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No